CLINICAL TRIAL: NCT03503123
Title: Deventilation Dyspnea in Patients With Chronic Obstructive Pulmonary Disease After Switching Off From Non-invasive Ventilation
Brief Title: Deventilation Dyspnea in COPD Patients Using NIV
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Marieke Duiverman, Post-doc, Pulmonary physician, University Medical Center Groningen
Other Study IDs: 201800263
Record Dates: First submitted 2018-04-09; First posted 2018-04-19 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: COPD; Dyspnea; Mechanical Ventilation Complication
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Electromyography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients with deventilation dyspnoea: Ten severe COPD patients (age>18yr) using chronic NIV with severe symptoms of deventilation dyspnoea (Borg Dyspnoea Scale ≥ 5)
  Interventions: Device: Monitoring physiology with Electrical Impedance Tomography, Electromyography and transcutaneous carbon dioxide measurements.
- COPD patients without deventilation dyspnoea: Ten severe COPD patients (age>18yr) using chronic NIV without symptoms of deventilation dyspnoea, matched with the first cohort/group with regard to the degree of static lung hyperinflation and NIV settings.
  Interventions: Device: Monitoring physiology with Electrical Impedance Tomography, Electromyography and transcutaneous carbon dioxide measurements.

INTERVENTIONS:
Device: Monitoring physiology with Electrical Impedance Tomography, Electromyography and transcutaneous carbon dioxide measurements. — Both groups get the same exposures: with measure physiology in both groups by using non-invasive measurement techniques. The techniques we use are Electrical Impedance Tomography to determine degree of hyperinflation. We use Electromyography to analyse respiratory drive. We measure transcutaneous carbon dioxide to assess the effects of non-invasive ventilation. Thereby, we will perform lung function tests.

SUMMARY:
Non-invasive ventilation (NIV) has shown to be an effective therapy for patients with Chronic Obstructive Pulmonary Disease (COPD) with Chronic Hypercapnic Respiratory Failure (CHRF). However, these COPD patients often report severe dyspnoea after switching off from NIV therapy, which leads to discomfort and distress. Currently, it is not known what causes this deventilation dyspnoea and therefore a possible treatment to prevent deventilation dyspnoea is not available. This study investigates possible mechanisms underlying the phenomenon of deventilation dyspnoea in COPD patients by monitoring the effects of NIV on the patient during an afternoon sleep.

DETAILED DESCRIPTION:
Rationale: Non-invasive ventilation (NIV) has shown to be an effective therapy for patients with Chronic Obstructive Pulmonary Disease (COPD) with Chronic Hypercapnic Respiratory Failure (CHRF). However, these COPD patients often report severe dyspnoea after switching off from NIV therapy, which leads to discomfort and distress. Currently, it is not known what causes this deventilation dyspnoea and therefore a possible treatment to prevent deventilation dyspnoea is not available.

Objective: 1) To investigate what mechanisms underlie the phenomenon of deventilation dyspnoea in COPD patients. 2) To investigate how the change in electrical impedance, measured with electrical impedance tomography (EIT), is related to the change in inspiratory capacity (IC) before and after sleep.

Study design: This study is an observational cohort study analysing changes occurring due to NIV which could explain the existence of deventilation dyspnoea in certain COPD patients using NIV. Ten patients with and ten patients without deventilation dyspnoea will visit the hospital for an afternoon sleep, during and after which several non-invasive measurements are performed to analyse the changes occurring during and after switching off NIV. In order to investigate the deventilation problem, we will measure:

1. the degree of hyperinflation due to NIV: this will be assessed by measuring the change in end-expiratory lung volume (EELV) with EIT before, during and after NIV, and the change in IC before and after sleeping with NIV.
2. the reduction of respiratory muscle activity due to NIV: this will be assessed by the change in electromyography of the frontal diaphragm before, during and after NIV.
3. the effectiveness of NIV in reducing CO2 level: this will be assessed with transcutaneous CO2 measurements (PtcCO2) before, during and after NIV.
4. the degree of deventilation dyspnoea before and after the afternoon sleep: this will be assessed with a 10-point Borg Scale.

Study population: Twenty severe COPD patients (age>18yr) using chronic NIV will be included in the study: 10 patients with severe symptoms of deventilation dyspnoea (Borg Dyspnoea Scale ≥ 5) and 10 patients without symptoms of deventilation dyspnoea, matched with regard to the degree of static lung hyperinflation and NIV settings.

Main study parameters/endpoints: Knowledge about the changes occurring during NIV in patients with COPD with deventilation dyspnoea. The percent change in EELV, IC, respiratory muscle activity and PtcCO2 will be calculated for both groups and correlated with the degree of deventilation dyspnoea.

ELIGIBILITY:
Inclusion Criteria:

* COPD with a NIV indication using chronic NIV
* Age > 18 years
* With or without deventilation dyspnea when switching off from NIV (depending on group/cohort)
* Written informed consent is obtained

Exclusion Criteria:

* COPD exacerbation within 2 weeks preceding the study
* Modification of ventilation within 2 weeks preceding the study
* Having a poor compliance with NIV (usage of <4 h/day)
* Having other disorders leading to respiratory failure (such as morbid obesity, kyphoscoliosis, neuromuscular diseases, tuberculosis)
* Not being able to sleep 1.5 hour in the afternoon
* Having spinal injury, BMI>50, damaged or inflamed skin around the thorax or a cardiac pacemaker or other implanted devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the University Medical Center Groningen (UMCG). There is a large population of COPD patients using NIV known at the Home Mechanical Ventilation (HMV) Centre (around 120 patients). The pulmonologists know already at least 10 patients who suffer extremely from deventilation dyspnoea, which could possibly participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
End-expiratory lung volume | Through study completion, which is one day of NIV use. Compare the primary outcome before and after the afternoon sleep.
  The change in end-expiratory lung volume due to NIV-usage
Inspiratory capacity | Through study completion, which is one day of NIV use. Compare the primary outcome before and after the afternoon sleep.
  The change in inspiratory capacity due to NIV-usage
Respiratory muscle activity | Through study completion, which is one day of NIV use. Compare the primary outcome before and after the afternoon sleep.
  The change in respiratory muscle activity due to NIV-usage
Transcutaneous carbon dioxide | Through study completion, which is one day of NIV use. Compare the primary outcome before and after the afternoon sleep.
  The change in transcutaneous carbon dioxide due to NIV-usage

SECONDARY OUTCOMES:
Correlation of inspiratory capacity with end-expiratory lung volume | Through study completion, which is one day of NIV use. Compare the primary outcome before and after the afternoon sleep.
  To validate Electrical Impedance Tomography measurements to determine end-expiratory lung volume, we will compare these outcomes with the golden standard inspiratory capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pulmonary diseases, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No